CLINICAL TRIAL: NCT05415007
Title: Brief Intervention to Reduce Anxiety and Promote Resilience in Caregivers of Youth With Cancer
Brief Title: GOLD: Brief Intervention to Reduce Anxiety and Promote Resilience in Families of Youth With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-54525; PEDSVAR0063 (Other: OnCore); NCI-2023-00703 (Registry Identifier: National Cancer Institute: Clinical Trials Reporting Program)
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Any types of cancer
MeSH Terms: conditions — Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOLD Psychosocial Program (Experimental): Participant will receive a 2-hour interventional session. Its content will consist of two modules: (1) psychoeducation and coping, providing information in content areas such as side effects of cancer treatments, fever protocols, role disruption and (2) stress, triggers, and self care, where caregivers will be briefed on symptoms of and reactions to traumatic stress in order to help parents accurately label thoughts and emotions related to their child's cancer diagnosis.
  Interventions: Behavioral: GOLD Program
- Treatment-as-Usual (TAU) (Active Comparator)
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: GOLD Program — Participant will receive a 2-hour interventional session
  Arms: GOLD Psychosocial Program
Behavioral: Treatment as usual (TAU) — Participant will receive treatment-As-Usual which consist of information about diagnosis routinely-disseminated by personnel and providers.
  Arms: Treatment-as-Usual (TAU)

SUMMARY:
The purpose of this study is to examine a psychotherapeutic and psycho-educational intervention offered in virtual settings to caregivers of youth with cancer. Human subjects must be used because they are the object of the intervention.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE(S)- To examine the feasibility and accessibility of a brief intervention for caregivers of youth with newly-diagnosed cancer as a preliminary, data-generating step toward applying for a larger NCI R34 grant evaluating the efficacy of the program in a randomized controlled trial.

SECONDARY OBJECTIVE(S)- We hope to learn whether a psycho-educational, psychotherapeutic intervention offered in a virtual setting to caregivers of children diagnosed with cancer is feasible, is acceptable, and can prevent, minimize, or improve symptoms of psychological distress (including symptoms of anxiety, depression, and post-traumatic stress disorder). We also hope to further our understanding of family stress and expand the idea for a need of mental health services in pediatric oncology. We aim to further understand intervention strategies for domains of family stress, reducing levels of caregiver anxiety, and promoting resilience for caregivers. This is important because these symptoms can affect the quality of life of caregivers and affect their ability to adhere to their children's treatments.

ELIGIBILITY:
Inclusion and Exclusion Criteria: Parents

Inclusion

* Child (0-17yrs) with recent (<12 mo) cancer diagnosis
* Fluent in English
* Consent to research

Exclusion:

* Lack of proficiency in written and spoken English
* Parent is under age 18
* Active Suicidal Ideation
* Child with cancer does not provide assent

Inclusion and Exclusion Criteria: Children

Inclusion:

* Recent (<12 mo) cancer diagnosis in child
* 8-17 Years old
* Provides assent to participate in the study

Exclusion:

* Cannot read English
* Parent is not enrolled in the study

Anyone who is not a caregiver of children who have been diagnosed with cancer within the past 12 months will be excluded.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of caregivers who enroll in the GOLD program | 1 month
  Measurement will be based on the percentage of caregivers who provide consent, and are retained in the program through 1-month follow-up.

SECONDARY OUTCOMES:
Acceptability of the GOLD Program for caregivers | 1 month
  Acceptability will be measure by the percentage of caregivers who provide complete data, and who are retained through 1-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Victoria E. Cosgrove, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Institute, San Francisco, California, United States